CLINICAL TRIAL: NCT04945785
Title: " SAVE Study (Switch AdVagraf® to Envarsus®) for Fast Metabolizers Kidney Transplant Recipients"
Acronym: SAVE
Status: Active, not recruiting | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC20_0443
Record Dates: First submitted 2021-06-01; First posted 2021-06-30 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Renal Transplant Failure

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- control: Before switch Advagraf to Envarsus
  Interventions: Other: No intervention
- case: After switch Advagraf to Envarsus
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — no intervention

SUMMARY:
The use of calcineurin inhibitors (CNIs) in kidney transplantation is the gold standard treatment to prevent episodes of rejection. Nevertheless, CNIs have side effects and are in particular nephrotoxic for the kidney transplant. Monitoring CNI dosages is fundamental for the clinician, in order to find the right balance between toxicity and prevention of rejection. Several recent studies suggest that a Radio Residual Concentration / Dosage (C0 / D) less than 1.05 (patients with rapid metabolizers) is associated with poor graft function (eGFR) and decreased kidney transplant survival. LCPT prolonged-release tacrolimus (Novel Once-Daily Extended-Release Tacrolimus. Prolonged-release tacrolimus: Envarsus®) is a marketed form of tacrolimus with interesting pharmacokinetic properties: daily intake, reduction of the absorption peak (Meltodose® technology ) and reduction of the total CNI dose by 30% to obtain an equivalent CO compared to other molecules on the market (Advagraf®, Prograf®). Thus, the use of LCPT in patients rapid metabolisers in relay of Advagraf® or Prograf® could make it possible to decrease renal toxicity while preserving rejection, by increasing the C0 / D ratio.

The investigators propose a pilot study aiming to study a prospective cohort of rapid metabolisers patients put on Envarsus at one month of transplant compared to a historical cohort, in terms of C0 / D ratio, function and survival of the renal graft.

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥ 18 years old
* 1st or 2nd kidney transplant
* Transplantation from a deceased donor (Encephalic death or arrested heart Maastricht III) or living donor
* C0 / D ratio <1.05 at one month of kidney transplant
* Renal graft function <60ml / min (eGFR estimate by CKD-EPI or MDRD).

Exclusion Criteria:

* Patient ≤ 18 years old, under guardianship or protected
* Graft rank ≥ 3
* Renal graft function <30 ml / min (eGFR estimate by CKD-EPI or MDRD)
* Presence of pre-transplant DSA (threshold> 2000 MFI)
* Occurrence of histologically proven rejection during the 1st month of transplant
* Presence of another functional transplant (heart / lung / liver / pancreas) or kidney bi-transplant
* Transplantation from a living donor
* Transplantation from an arrested heart donor Maastricht II

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Major patients with row 1 or 2 renal transplants (1st or 2nd transplant) rapid metabolizers defined by a C0 / D ratio <1.05 at one month post transplant, with impaired function of the graft. 75 patients will be prospectively included in the Advagraf® or Prograf® switch cohort for Envarsus® during their renal transplant follow-up. 150 patients matched on age, graft rank, type of donor (standard criteria / expanded criteria) and C0 / D at one month of grafting will constitute the retrospective control cohort extracted from the database in Nantes.
Sampling Method: Probability Sample
Enrollment: 226 (Actual)
Dates: Start 2021-07-28 (Actual); Primary Completion 2025-05-28 (Actual); Study Completion 2026-05-28 (Estimated)

PRIMARY OUTCOMES:
Improvement of kidney allograft between month 1 and month 12 | 12 months
  comparison of eGFR (estimated Glomerular Filtration Rate) level at M12 by using the MDRD formula between Envarsus® and Advagraf® groups.

CONTACTS AND LOCATIONS:
Overall Officials: Jacques DANTAL, Principal Investigator — Nantes University Hospital
Locations (1):
- CHU de Nantes, Nantes, France

IPD SHARING:
Plan to Share IPD: Undecided